CLINICAL TRIAL: NCT01687595
Title: A Phase 2a, Multicenter, Double-blinded, Randomized, 2-Period Trial to Evaluate the Effect of HerpV Administered in Combination With the Stimulon® Adjuvant QS-21 on Viral Shedding in Adults With Recurrent Genital Herpes
Brief Title: Biological Efficacy Study of HerpV Vaccine With QS-21 to Treat Participants With Recurrent Genital Herpes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-400-02
Record Dates: First submitted 2012-09-12; First posted 2012-09-19 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Herpes Simplex Type 2
Keywords: herpes simplex virus type 2,; genital herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — saponin QA-21V1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HerpV 240 μg + QS-21 50 μg (Experimental): Participants will receive a combination of HerpV 240 micrograms (μg) and QS-21 50 μg injection subcutaneously at Weeks 0, 2 and 4 in treatment period 1. At Week 24, participants who completed treatment period 1 will receive a booster dose of combination of HerpV 240 μg and QS-21 50 μg in treatment period 2. Each treatment period will be followed by a washout period of 1 week.
  Interventions: Drug: HerpV and QS-21
- Placebo (Placebo Comparator): Participants will receive a placebo injection subcutaneously at Weeks 0, 2 and 4 in treatment period 1 and at Week 24 in treatment period 2. Each treatment period will be followed by a washout period of 1 week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HerpV and QS-21 — HerpV (recombinant human heat shock protein 70 [rh-Hsc70] polyvalent peptide complex) in combination with adjuvant QS-21
  Other Names: AG-707
  Arms: HerpV 240 μg + QS-21 50 μg
Drug: Placebo — phosphate buffered saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of recombinant human heat shock protein 70-polyvalent peptide complex (HerpV) vaccine administration on recurring episodes of genital herpes by evaluating viral shedding before and after treatment.

DETAILED DESCRIPTION:
This study will evaluate the biological effectiveness and safety of the HerpV vaccine in combination with adjuvant QS-21. The Safety and tolerability of HerpV plus QS-21 will also be evaluated by collecting number and severity of adverse events throughout the study.

Participants will undergo a baseline/ screening period. This is a 45 day period when the participant collects a swab of the genital area each day. In case of a recurrence, participant will be required to collect two swabs a day. If the participant collects at least 80% of the swabbing samples and meets all eligibility criteria they may enroll in the study.

Study Period 1 consists of three treatments and a 45 day swabbing period after the last treatment. The participant will collect swabs of the genital region each day for 45 days.

Participants who successfully complete Study Period 1 will proceed to Study Period 2. They will receive a booster injection of study drug or placebo according to their original randomization assignment. The participants will again enter a 45 day swabbing period, collecting swabs of the genital area each day for 45 days.

ELIGIBILITY:
Inclusion Criteria:

* Seropositive for herpes simplex virus type 2 (HSV-2)
* Clinically active genital herpes defined as a history of 1-9 episodes per year for at least 1 year prior to screening or 1 year prior to beginning suppressive therapy.
* Willing to either use an effective method of contraception or abstain from sexual intercourse throughout the 48-week study period.
* If female of childbearing potential, have a negative serum pregnancy test.
* Agree to not receive any other investigational drugs while enrolled in this study.
* The above criteria must be met before participants are allowed to enter the 45-day swabbing period to be screen for the study.
* Completion and collection of greater than or equal to 80% (36 days) of the 45-day consecutive daily genital swabs.

Exclusion Criteria:

* Severe active infection, compromised cardiopulmonary function, or other serious medical illness that, in the opinion of the principal investigator, would prevent study completion.
* A history of herpes simplex virus (HSV) infection of the eye (herpes simplex interstitial keratitis or uveitis), or herpes-associated erythema multiforme.
* A history of immune suppression or autoimmune disorder.
* Continued use of suppressive anti-viral therapy for HSV-2; a 1 week washout of any anti-viral therapy (suppressive and episodic) is required prior to initiating the swabbing period.
* Concomitant use of systemic corticosteroids or immune-suppressive medications. The use of nasal steroids is acceptable.
* Human immunodeficiency virus (HIV) positive.
* Presence of active Hepatitis B or C infection.
* Known hypersensitivity or allergies to acyclovir or valacyclovir.
* Pregnant or breast-feeding women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agenus Medical Monitor, Study Director — Agenus Inc.
Locations (5):
- United States (5):
  - Westover Heights Clinic, Portland, Oregon
  - Center for Clinical Studies - Texas Medical Center, Houston, Texas
  - Center for Clinical Studies - Cypress, Houston, Texas
  - Center for Clinical Studies- Webster, Houston, Texas
  - University of Washington Virology Research Clinic, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wald A, Koelle DM, Fife K, Warren T, Leclair K, Chicz RM, Monks S, Levey DL, Musselli C, Srivastava PK. Safety and immunogenicity of long HSV-2 peptides complexed with rhHsc70 in HSV-2 seropositive persons. Vaccine. 2011 Nov 3;29(47):8520-9. doi: 10.1016/j.vaccine.2011.09.046. Epub 2011 Sep 21. PMID 21945262

RESULTS

PARTICIPANT FLOW:
Groups:
- HerpV + QS-21: Participants received a combination of HerpV (recombinant human heat shock protein 70 [rh-Hsc70] polyvalent peptide complex) 240 micrograms (μg) and QS-21 50 μg injection subcutaneously at Weeks 0, 2 and 4 in treatment period 1. At Week 24, participants who completed treatment period 1 received a booster dose of combination of HerpV 240 μg and QS-21 50 μg in treatment period 2. Each treatment period was followed by a washout period of 1 week.
- Placebo: Participants received placebo (phosphate buffered saline [PBS]) injection subcutaneously at Weeks 0, 2 and 4 in treatment period 1 and at Week 24 in treatment period 2. Each treatment period was followed by a washout period of 1 week.
Period: Overall Study
Arm/Group | HerpV + QS-21 | Placebo
Started | 70 | 10
Received at Least 1 Dose of Study Drug | 70 | 10
Completed | 0 | 0
Not Completed | 70 | 10
Not completed — Withdrawal by Subject | 8 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Investigator's decision | 1 | 0
Not completed — Sponsor's decision | 1 | 0
Not completed — Noncompliance | 1 | 2
Not completed — Other than specified | 56 | 7

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study medication according to initial randomization.
Groups:
- HerpV + QS-21: Participants received a combination of HerpV 240 μg and QS-21 50 μg injection subcutaneously at Weeks 0, 2 and 4 in treatment period 1. At Week 24, participants who completed treatment period 1 received a booster dose of combination of HerpV 240 μg and QS-21 50 μg in treatment period 2. Each treatment period was followed by a washout period of 1 week.
- Placebo: Participants received placebo (PBS) injection subcutaneously at Weeks 0, 2 and 4 in treatment period 1 and at Week 24 in treatment period 2. Each treatment period was followed by a washout period of 1 week.
- Total: Total of all reporting groups
Arm/Group | HerpV + QS-21 | Placebo | Total
Number analyzed (Participants) | 70 | 10 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (8.00) | 33.7 (6.22) | 35.6 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 6 | 48
  Male | 28 | 4 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Overall Viral Shedding Rate From Baseline (Week -7 to 0) to Post-treatment Period (Weeks 6 to 13)
Description: The viral shedding rate was defined as the number of days with genital swab positive for herpes simplex virus (HSV) deoxyribonucleic acid (DNA), as measured by quantitative real-time polymerase chain reaction (PCR), relative to the total number of days with available swabs.
  The viral shedding rate was defined as the number of days with genital swab positive for herpes simplex virus (HSV) deoxyribonucleic acid (DNA), as measured by quantitative real-time polymerase chain reaction (PCR), relative to the total number of days with available swabs. Overall viral shedding rate = number of days with positive PCR/total number of days PCR results collected. Change in overall viral shedding rate was calculated within participants comparing baseline with post-treatment, and summarized across all participants.
  Percent change in viral shedding rate and 95% CI are reported.
Time Frame: Baseline, Weeks 6-13
Population: Efficacy population included all randomized participants who received all 3 vaccinations of Herp-V vaccine and were compliant with the study procedures. This outcome measure was planned to be analyzed for "HerpV + QS-21" arm only.
Measure: Number (95% Confidence Interval); unit: percentage change
Arm/Group | HerpV + QS-21
Number analyzed (Participants) | 70
percentage change | 13.53 [2.38 to 23.40]

2. Primary Outcome: Percent Change in Overall Viral Shedding Rate From Baseline (Week -7 to 0) to Post-treatment Period (Weeks 26 to 33)
Description: The viral shedding rate was defined as the number of days with genital swab positive for HSV DNA, as measured by quantitative real-time PCR, relative to the total number of days with available swabs.
  The viral shedding rate was defined as the number of days with genital swab positive for herpes simplex virus (HSV) deoxyribonucleic acid (DNA), as measured by quantitative real-time polymerase chain reaction (PCR), relative to the total number of days with available swabs. Overall viral shedding rate = number of days with positive PCR/total number of days PCR results collected. Change in overall viral shedding rate was calculated within participants comparing baseline with post-treatment, and summarized across all participants.
  Percent change in viral shedding rate and 95% CI are reported.
Time Frame: Baseline, Weeks 26-33
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage change
Arm/Group | HerpV + QS-21
Number analyzed (Participants) | 70
percentage change | 12.78 [0.83 to 23.28]

3. Other Pre Specified Outcome: Number of Participants With Peripheral Blood Mononuclear Cell Immune Response at Any Time
Time Frame: Baseline through Week 26
Population: Efficacy population included all randomized participants who received all 3 vaccinations of Herp-V vaccine and were compliant with the study procedures. Here, Overall number of participants analyzed signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | HerpV + QS-21 | Placebo
Number analyzed (Participants) | 61 | 8
Participants | 46 | 1

4. Other Pre Specified Outcome: Number of Participants With CD8+ Immune Response at Any Time
Time Frame: Baseline through Week 26
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HerpV + QS-21 | Placebo
Number analyzed (Participants) | 61 | 8
Participants | 32 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to Week 76
Description: Safety population included all randomized participants who received at least 1 dose of study medication according to initial randomization.
Arm/Group | HerpV + QS-21 | Placebo
Serious Adverse Events (participants affected / at risk) | 3/70 | 0/10
Other Adverse Events (participants affected / at risk) | 67/70 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HerpV + QS-21 (N=70) | Placebo (N=10)
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | HerpV + QS-21 (N=70) | Placebo (N=10)
Anemia (Blood and lymphatic system disorders) | 3 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Hyperacusis (Ear and labyrinth disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Erythema of eyelid (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Eyelid edema (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Abdominal pain, upper (Gastrointestinal disorders) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 25 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 30 | 6
Paresthesia, oral (Gastrointestinal disorders) | 2 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 1
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2
Asthenia (General disorders) | 1 | 0
Axillary pain (General disorders) | 1 | 0
Chills (General disorders) | 12 | 0
Fatigue (General disorders) | 57 | 6
Feeling cold (General disorders) | 1 | 0
Induration (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Influenza-like illness (General disorders) | 1 | 0
Injection-site cyst (General disorders) | 1 | 0
Injection-site erythema (General disorders) | 56 | 0
Injection-site hematoma (General disorders) | 6 | 1
Injection-site induration (General disorders) | 16 | 0
Injection-site pain (General disorders) | 66 | 5
Injection-site paresthesia (General disorders) | 0 | 1
Injection-site pruritus (General disorders) | 18 | 1
Injection-site rash (General disorders) | 2 | 0
Injection-site swelling (General disorders) | 42 | 0
Injection-site ulcer (General disorders) | 1 | 0
Injection-site vesicles (General disorders) | 1 | 0
Injection-site warmth (General disorders) | 4 | 0
Pyrexia (General disorders) | 11 | 0
Vaccination-site warmth (General disorders) | 1 | 0
Hypertransaminasemia (Hepatobiliary disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Chlamydial infection (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis, viral (Infections and infestations) | 3 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 4 | 0
Nasopharyngitis (Infections and infestations) | 7 | 0
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis, streptococcal (Infections and infestations) | 2 | 1
Rash, pustular (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 5 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Vaginal abscess (Infections and infestations) | 1/42 | 0/6 — This is a gender specific AE that affects only female participants.
Vulvovaginal candidiasis (Infections and infestations) | 0/42 | 1/6 — This is a gender specific AE that affects only female participants.
Vulvovaginitis (Infections and infestations) | 1/42 | 0/6 — This is a gender specific AE that affects only female participants.
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 2 | 1
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood growth hormone decreased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 56 | 4
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Breast cancer, in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer, stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 7 | 0
Headache (Nervous system disorders) | 49 | 7
Hyperesthesia (Nervous system disorders) | 2 | 0
Nerve compression (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 2 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Mid-cycle spotting (Reproductive system and breast disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/42 | 0/6 — This is a gender specific AE that affects only female participants.
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 1
Bladder discomfort (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 1/42 | 0/6 — This is a gender specific AE that affects only female participants.
Menstrual disorder (Reproductive system and breast disorders) | 1/42 | 0/6 — This is a gender specific AE that affects only female participants.
Pelvic pain (Reproductive system and breast disorders) | 1/42 | 0/6 — This is a gender specific AE that affects only female participants.
Penile pain (Reproductive system and breast disorders) | 1/28 | 0/4 — This is a gender specific AE that affects only male participants.
Sexual dysfunction (Reproductive system and breast disorders) | 1 | 0
Vaginal laceration (Reproductive system and breast disorders) | 1/42 | 0/6 — This is a gender specific AE that affects only female participants.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis, contact (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema, multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritis, generalized (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash, pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes